CLINICAL TRIAL: NCT00048893
Title: A Multicenter Phase I-II Study of Tumor Vaccine Following Chemotherapy in Patients With Metastatic Breast Cancer Untreated With Chemo/Radiation in the Previous 18 Months: Vaccine-Induced Bias of T-Cell Repertoire Reconstitution After T-Cell Re-Infusion
Brief Title: Vaccine and Chemotherapy for Previously Untreated Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was closed to accrual due to very poor enrollment.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Claude Sportes, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030040; 03-C-0040; NCT00053170 (obsolete NCT alias)
Record Dates: First submitted 2002-11-08; First posted 2002-11-11 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-03

CONDITIONS: Breast Neoplasms; Metastases, Neoplasm
Keywords: CEA vaccine; Metastatic Breast Cancer; T- Cell Repertoire; High-dose Chemotherapy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Filgrastim; sargramostim; Colony-Stimulating Factors; Cyclophosphamide; Doxorubicin; fludarabine phosphate; Paclitaxel; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: recombinant fowlpox-CEA(6D)/TRICOM vaccine — 4 x 10^8 pfu given monthly subcutaneously for three doses in the first series and three doses on each of the intermediate and late re-immunizations (total 9 doses).
Biological: recombinant vaccinia-CEA(6D)/TRICOM vaccine — rV-CEA (6D)/Tricom concomitantly with sargramostim (rGM-CSF). 1.2 x 10^8 pfu x 1 dose subcutaneously.
Biological: filgrastim — 5 mcg/kg/day subcutaneously
  Other Names: Neupogen
Biological: sargramostim — 100 mcg daily for 4 consecutive days at the same site as the rF-CEA (6D)/Tricom vaccine. The first dose will be given with the vaccine.
  Other Names: rGM-CSF; Leukine
Drug: cyclophosphamide — First induction chemotherapy: 2700 mg/m^2 per cycle (900 mg/m^2 per day intravenous over 1 hour for 3 consecutive days, days 1-3).
  Second induction: 600 mg/m^2 per cycle (600 mg/m^2 intravenous over 1 hour day 1.
  Immune depleting chemotherapy: 2400 mg/m^2 per cycle (600 mg/m^2 per day intravenous over 1 hour for 4 consecutive days, days 1-4).
  Other Names: Cytoxan
Drug: doxorubicin hydrochloride — 60 mg/m^2 per cycle (60 mg/m^2 slow intravenous push day 1).
  Other Names: Adriamycin
Drug: fludarabine phosphate — 120 mg/m^2 (30 mg/m^2 per day intravenous over 30 minutes for 4 consecutive days (days 1-4)).
  Other Names: Fludara
Drug: paclitaxel — 160 mg/m^2 per cycle (53.3 mg/m^2 per day by continuous intravenous infusion over 24 hours for 3 consecutive days 1-3).
  Other Names: Taxol
Drug: Mesna — Percent equals fraction of total daily cyclophosphamide dose. Initial: 20% of cyclophosphamide dose given intravenously (IV) mixed with cyclophosphamide.
  3 hours post completion of cyclophosphamide: 20% intravenously (IV) or 40% by mouth (PO) 6 hours post completion of cyclophosphamide: 20% intravenously (IV) or 40% by mouth (PO) 9 hours post completion of cyclophosphamide: 20% intravenously (IV) or 40% by mouth (PO)
  Other Names: Mesnex

SUMMARY:
This study will evaluate the effectiveness of chemotherapy and a combination of vaccines to treat metastatic breast cancer (breast cancer that has spread beyond the breast) in patients whose cancer cells have a protein called carcinoembryonic antigen (CEA) on their surface. Patients who require surgery or radiation therapy, or both, will receive these treatments as well.

Patients 18 years of age and older with previously untreated metastatic breast cancer may be eligible for this study. Newly diagnosed patients may not have received prior chemotherapy. Patients previously diagnosed with local disease may have received chemotherapy or radiation therapy at least 18 months before entering the current study. Patients may have received hormonal therapy for stage IV disease. Candidates are screened with a medical history and physical examination, blood and urine tests, x-rays, heart and lung tests, and a test to determine the presence of CEA on their tumor cells.

Participants undergo the following procedures:

1. Central venous line: Under local or general anesthesia, an intravenous catheter (plastic tube) is inserted into a major vein in the chest. It is used to give chemotherapy and other medications and to withdraw blood samples.
2. Apheresis: Before beginning treatment and at various times before and after chemotherapy, patients undergo apheresis to collect white blood cells for later re-infusion at the time of immunizations and to evaluate the body's response to the vaccines. For this procedure, blood is collected through the central venous catheter and circulated through a machine that separates the white cells from the rest of the blood. The white cells are removed and frozen for later use. The rest of the blood is returned to the patient through the catheter.
3. First vaccine: Before starting chemotherapy, patients receive one subcutaneous (under the skin) injection of a vaccine called rV-CEA-Tricom, along with subcutaneous injections of granulocyte macrophage colony stimulating factor (GM-CSF) (Sargramostim), a drug that stimulates the bone marrow to release white blood cells and white cell precursors into the bloodstream.
4. Chemotherapy:

   * Taxol (paclitaxel)/Cytoxan (cyclophosphamide): Patients receive three to five cycles of Taxol and Cytoxan. Taxol is given as a continuous 72-hour intravenous (intravenous (IV), through a vein) infusion and Cytoxan is given daily for 3 days, intravenously, over 1 hour. Cycles are 21 to 42 (usually 28) days. After each cycle, patients also receive growth colony stimulating factor (G-CSF) (a drug that helps boost white cells.

DETAILED DESCRIPTION:
BACKGROUND: Metastatic breast cancer remains to this day a mostly incurable disease, with less than 10% of patients reaching a long-term disease free survival. This study proposes using an immune-depleting chemotherapy as platform for immunotherapy. It is based on the following hypotheses and understanding:

* The combination of dose-intensive followed by immune-depleting chemotherapy provides a platform for subsequent immunotherapy by:

  1. Lengthening the progression-free survival period, thus allowing time for a slow acting therapy such as vaccination to be effective.
  2. Maximally decreasing the patient's tumor burden. This has been shown both in clinical and experimental settings to be desirable if not necessary for immunotherapy to be effective.
  3. Decreasing the tumor burden which may also decrease a tumor-induced immuno-suppressive effect linked to tumor bulk.
  4. Providing tumor antigen exposure following immune depletion in the form of repeated immunizations. This may take advantage of the pattern of immune reconstitution following immune depleting therapy at early time points (antigen-driven peripheral expansion of T-cells) and the renewal of a T-cell repertoire biased towards tumor antigens and anti-tumor responses at later time points.
* Low antigenicity of tumor antigens and immune tolerance may be overcome in a clinically relevant fashion by providing exposure to the tumor antigens (the carcino-embryonic antigen CEA) in a more immunogenic presentation along with added co-stimulatory signal (in the form of two poxvirus-based recombinant vaccines).
* Due to the post immune depletion defects and delay in immune reconstitution, an adequate immune response to vaccines may not occur unless the patients are provided, following immune depletion, with unaltered T-cells in the form of re-infusion of pre-chemotherapy lymphocytes.

The late recovery of thymic function (18 to 24 months) with reappearance of naive T-cells may play a determinant role in the prevention of later disease progression. It is the rationale for a late series of immunizations.

ELIGIBILITY: Patients with metastatic breast cancer untreated with chemotherapy or radiation in the previous 18 months with CEA positivity in either the tumor or the serum.

OBJECTIVES: The primary objectives are to evaluate biologically this immunization strategy by assessing CEA specific T-cell responses as well as clinically by comparing the patient event free survival (EFS) to our historical control (protocol 96-C-0104) in which patients have received the same conventional therapy but no immunization

DESIGN: Before any chemotherapy patients will be immunized with one of two tumor-specific, recombinant, poxvirus-based deoxyribonucleic acid (DNA) Tricom vaccines and sensitized lymphocytes will be cryopreserved. Patients will then receive conventional induction therapy with Paclitaxel, Cyclophosphamide and Doxorubicin, surgery and / or radiation as indicated for local control, then immune depleting chemotherapy with Fludarabine & Cyclophosphamide. Following immune depletion, patients will receive 9 immunization boosts over the next 30 months. Patients whose disease progress through the vaccination schedule, may, under certain circumstances, receive further vaccinations under a more intensive schedule (monthly).

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients must have a diagnosis of metastatic infiltrating carcinoma of the breast including hormone receptor testing. At least one site of metastatic disease must have been confirmed by pathologic or cytologic material. In the choice of a biopsy site, the PI will weigh the morbidity the diagnostic procedure against the probability of positive yield of the diagnostic procedure.

All pathologic material must be reviewed by the Pathology Laboratory of the National Cancer Institute (NCI) before treatment.

The tumor MUST stain positive for CEA, by standard immuno-histochemistry performed at the Pathology Laboratory of the NCI.

--Method: 5 microM formalin-fixed paraffin-embedded sections are deparaffinized and blocked with methanol-30% hydrogen peroxide (H2O2). After antigen retrieval by boiling in citrate buffer, or heating in a microwave oven for 10 minutes, slides are incubated with monoclonal antibodies anti-CEA (diluted 1/1000 Dako). Then, slides are immunostained with avidin-biotin-peroxidase complex and developed with diaminobenzidine. Harris' hematoxylin was used to counter stain the slides. Positivity is defined as greater than 30% of cells staining.

Patients may be newly diagnosed with metastatic breast carcinoma or known to have breast carcinoma.

* If newly diagnosed, patients may not have received any chemotherapy for this disease before entry on study.
* If previously treated for breast cancer, patients may have received chemotherapy or radiation as adjuvant treatment for non-metastatic disease or metastatic disease but not in the previous 18 months.
* Patients may have been on hormonal therapy for stage IV disease. Patients with disease progression on hormonal therapy alone are eligible.

Karnofsky performance status of greater than or equal to 70% (Eastern Cooperative Oncology Group (ECOG) 0 or 1)

Ejection fraction by multi-gated acquisition scan (MUGA) or 2-dimensional (2-D) echocardiogram within normal institutional limits. In case of insufficient ejection fraction, a stress echocardiogram will be performed. In case of an ejection fraction greater than 35 % but less than 45%, the patient will remain eligible for the study if the increase of ejection fraction with stress is estimated at 10% or more.

Creatinine clearance greater than or equal to 60 cc/min

Normal urinalysis; if proteinuria is present it must be quantified at less than 1 g / 24 h on a measured 24 h urine collection

Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 3 times the upper limit of normal except if believed to be due to tumor involvement of the liver prior to induction therapy.

Bilirubin less than 1.5 (except if due to tumor involvement prior to induction therapy or in cases of Gilbert's disease).

Absolute Neutrophil Count greater than l000 / mm^3 and Platelet count greater than 90,000

Corrected carbon monoxide diffusing capacity (DLCO) greater than 50%

No history of abnormal bleeding tendency or predisposition to repeated infections.

Patient must be able to avoid close contact with children under 3 years old, pregnant women, individuals with eczema or other skin conditions, and immuno-suppressed people for 2 weeks after initial vaccination. (see protocol for specific exclusion criteria for vaccinia administration). Patients must agree to make specific arrangements, if necessary, in order to comply and be eligible.

Patients must be able to give informed consent.

EXCLUSION CRITERIA:

Age less than 18 years

Patients in whom an urgent or emergent clinical situation does not safely allow for the short delay in initiating the Concurrent Therapy (as defined in protocol) necessary for the pre-treatment immunization and lymphocyte collection (at the discretion of the PI).

Patients requiring chronic immunosuppressive therapy (including corticosteroids) for any medical condition.

Patients with an autoimmune disease: autoimmune neutropenia, thrombocytopenia, or hemolytic anemia; Rheumatoid Arthritis, Systemic Lupus Erythematosus, Sjogren syndrome, Scleroderma, Systemic Sclerosis, Myasthenia Gravis; Multiple sclerosis, Goodpasture syndrome; Addison's disease, Hashimoto's thyroiditis, or active Graves' disease)

Any abnormality on the following tests suggestive of an autoimmune disease: anti-nuclear antibody (ANA), anti-deoxyribonucleic acid (DNA), triiodothyronine (T3), thyroxine (T4), thyroid stimulating hormone (TSH) after review with appropriate consultant. Patients with endocrine disease that is controlled by replacement therapy including, diabetes, thyroid and adrenal disease or vitiligo may be enrolled.

Patients with active inflammatory bowel disease

Patients with clinically significant cardiomyopathy requiring treatment or symptomatic congestive heart failure (CHF), symptomatic arrhythmia that is not controlled by medication, unstable coronary artery disease (CAD) such as unstable angina who require active intervention, and patients with a recent infarction or cerebrovascular accident (CVA) within the past 6 months

Patients testing positive for human immunodeficiency virus (HIV) or hepatitis B or C

Patients known or found to be pregnant or those unwilling to discontinue breastfeeding. The effects of the chemotherapy, vaccines, and the medications used in this study are highly likely to be harmful to a fetus. The effects upon breast milk are also unknown and may be harmful to the infant; therefore, women should not breastfeed while on this study.

Patients of childbearing age who are unwilling to practice an effective form of contraception. Patients of childbearing potential must use an effective method of contraception while they are on-study; effective methods include intrauterine device (IUD), hormonal (birth control pills, injections, or implants), tubal ligation/hysterectomy (self or partner), partner's vasectomy, or barrier methods (condom, diaphragm, or cervical cap), or abstinence.

Patients with brain metastases.

Patients with an active second malignancy (excluding treated skin cancers or carcinoma in-situ) will be ineligible.

Patients with a life expectancy reasonably estimated at less than 6 months.

Patients may be excluded at the discretion of the principal investigator (PI) if it is deemed that allowing participation would represent an unacceptable medical or psychiatric risk.

History of splenectomy

Allergy to eggs

Several exclusion criteria are specific to vaccinia administration:

The recombinant vaccinia vaccine should not be administered if the following apply to either recipients or, for at least two weeks after vaccination, to their close household contacts (Close household contacts are those who share housing or have close physical contact):

* Persons with active or a history of eczema or other eczematoid skin disorders
* Persons with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne or other open rashes or wounds) until condition resolves;
* Pregnant or nursing women
* Children under 3 years of age;
* Immunodeficient or immunosuppressed persons by disease or therapy, including HIV infection.
* History of seizures, encephalitis, or multiple sclerosis
* History of allergy or complications with past vaccinia vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2002-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Sportes, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey

REFERENCES:
- See also: Common Terminology Criteria for Adverse Events (CTCAE) — http://ctep.cancer.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- Carcinoembryonic Antigen (CEA)-Tricom Vaccines: (fV-CEA (6D)/Tricom with sargramostim (rGM-CSF) 1.5 x 10^8 plaque-forming unit (pfu) x 1 dose subcutaneously
Period: Overall Study
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 8
  White | 26
  Unknown or Not Reported | 2
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival as Measured by Clinical Evaluation and Tumor Measurements by Imaging
Description: Complete response (CR) is the complete disappearance of all measurable and evaluable disease. Partial response (PR) is a decrease of greater than or equal to 50% in the sum of the products of the longest perpendicular dimensions of all measurable target lesions. Stable disease (SD) is any decrease of less than 50% or increase less than 25% in the sum of the longest perpendicular dimensions of measurable disease. Progressive disease (PD) is a greater than 25% increase in the sum of the longest perpendicular dimensions of any measurable disease.
Time Frame: time to progression, response rate: evaluation every 3 months for 3 years, then every 6 months for one year (fourth year), then yearly thereafter until taken off study
Population: The study was closed to accrual due to very poor enrollment. No meaningful data analysis was possible on the small number of accrued subjects, so none was done.
Measure: Number; unit: Months
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 91 months
Measure: Number; unit: Participants
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Number analyzed (Participants) | 37
Participants | 11

3. Secondary Outcome: Log Change in Precursor Frequency as Measured by Elispot.
Description: The log change in CEA-specific T cell precursor frequency will be calculated between values obtained at baseline and 5 months post immune depletion. A change equal to 1.0 standard deviation (SD) of the log change is significant.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: log change in CEA-specific T cell precur
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Number analyzed (Participants) | 0

4. Secondary Outcome: Log Change of CD4 CEA-specific Immune Responses and Their Kinetics as a Surrogate Marker for Clinical Anti-tumor Activity of the Vaccines
Description: Response is evaluated by CD4 response to CEA soluble protein. The log change in precursor frequencies will be calculated between values obtained at baseline and five months post immune depletion. By flow cytometry of peripheral blood lymphocyte frequency of potential killer cells directed to the CEA protein.
Time Frame: Baseline and 5 months post immune depletion
Population: as for outcome 1
Measure: Number; unit: log change of CD4 CEA specific precursor
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Number analyzed (Participants) | 0

5. Secondary Outcome: Immune Response to the Vaccine in Those Patients With Late Recovery of Thymic Function
Description: It is expected that delayed administration of a vaccine will result in enhancement of immune response to the vaccine in those patients with later recovery of thymic function as evidenced by change in lymphocyte subsets in the blood.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: Cells/L
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Months of Progression Free Survival
Description: The time period a participant remains free from progressive disease. Progressive disease (PD) is defined as a greater than 25% increase in the sum of the longest perpendicular dimensions of any measurable disease or the appearance of new disease or an increase in evaluable disease.
Time Frame: After the immune depletion cycle
Population: as for outcome 1
Measure: Number; unit: Months
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With an Immune Response as a Result of the Salvage Immunization Schedule
Description: Patients showing disease progression or recurrence at any point after the start of the early immunizations series may continue on study in accordance to the off study criteria and will be receiving monthly rF immunizations for a total of 12 months or until further disease progression meets the off study criteria. Immune response as evidenced by change in lymphocyte subsets in the blood.
Time Frame: 6 weeks, than 6, 12, 18, 24, 30, 36 (3y), 42, 48 (4y), 60 and 72 months after completion of immune chemotherapy
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With a Clinical Response
Description: Defined as measurable disease (any solid lesion that can be measured accurately in at least one dimension), evaluable disease (disease not readily measurable but can be clinically assessed), complete response (complete disappearance of all measurable and evaluable disease), partial response (decrease of greater than or equal to 50%), stable disease (any decrease of less than 50% or increase less than 25% in the sum of the longest perpendicular dimensions), or progressive disease (greater than 25% increase in the sum of the longest perpendicular dimensions of any measurable disease).
Time Frame: At the beginning of each cycle of chemotherapy (every 4 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 91 months
Arm/Group | Carcinoembryonic Antigen (CEA)-Tricom Vaccines
Serious Adverse Events (participants affected / at risk) | 11/37
Other Adverse Events (participants affected / at risk) | 11/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carcinoembryonic Antigen (CEA)-Tricom Vaccines (N=37)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (7)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Thrombosis/embolism (Cardiac disorders) | 1 (1)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 (1)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 1 (1)
Prothrombin time (PT) (Blood and lymphatic system disorders) | 2 (2)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0x10e9/L) (General disorders) | 5 (7)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase (Hepatobiliary disorders) | 1 (1)
Bilirubin (Hepatobiliary disorders) | 2 (4)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 1 (1)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 1 (1)
Catheter-related infection (Infections and infestations) | 5 (7)
Febrile neutropenia (Infections and infestations) | 8 (13) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0x10e9/L, fever>=38.5 degrees C)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e (Infections and infestations) | 2 (3)
Infection without neutropenia (Infections and infestations) | 2 (2)
Infection/Febrile Neutropenia-Other (Specify, infection:catheter-related infection) (Infections and infestations) | 1 (1)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Confusion (Nervous system disorders) | 1 (1)
Dizziness/lightheadedness (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carcinoembryonic Antigen (CEA)-Tricom Vaccines (N=37)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4 (4)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 4 (4)
Allergy-Other (Specify, itching & red splotches due to shellfish) (Immune system disorders) | 1 (1)
Autoimmune reaction (Immune system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 10 (172)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 10 (169)
Lymphopenia (Blood and lymphatic system disorders) | 10 (70)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 10 (118)
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 10 (11)
Transfusion: Platelets (Blood and lymphatic system disorders) | 5 (11)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 7 (23)
Edema (General disorders) | 3 (3)
Hypotension (General disorders) | 3 (3)
Phlebitis (superficial) (General disorders) | 2 (2)
Fibrinogen (Investigations) | 1 (1)
Partial thromboplastin time (PTT) (Investigations) | 6 (11)
Prothrombin time (PT) (Investigations) | 2 (3)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 8 (31)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0x10e9/L) (General disorders) | 7 (12)
Rigors, chills (General disorders) | 6 (11)
Sweating (diaphoresis) (General disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Flushing (Skin and subcutaneous tissue disorders) | 2 (2)
Injection site reaction (Skin and subcutaneous tissue disorders) | 10 (35)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 2 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1)
Wound-infectious (Skin and subcutaneous tissue disorders) | 1 (1)
Endocrine-Other (Specify,endocrine-other: hyperthyroid) (Endocrine disorders) | 2 (3)
Hot flashes/flushes (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 1 (2)
Anorexia (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 7 (15)
Dyspepsia/heartburn (Gastrointestinal disorders) | 3 (6)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 4 (7)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal-Other (Specify,gastrointestinal:hemorrhoid; indigestion) (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (19)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 8 (12)
Vomiting (Gastrointestinal disorders) | 5 (12)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Hematuria (in the absence of vaginal bleeding) (Blood and lymphatic system disorders) | 5 (13)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 2 (2)
Alkaline phosphatase (Hepatobiliary disorders) | 5 (11)
Bilirubin (Hepatobiliary disorders) | 5 (11)
Hepatic-Other (Specify, albumin_serum low) (Hepatobiliary disorders) | 2 (2)
Hypoalbuminemia (Hepatobiliary disorders) | 9 (56)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Blood and lymphatic system disorders) | 10 (36)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 9 (36)
Catheter-related infection (Infections and infestations) | 2 (2)
Febrile neutropenia (Infections and infestations) | 2 (2) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC<1.0x10e9/L, fever>=38.5 degrees C)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC<1.0x10e9/L (Infections and infestations) | 3 (8)
Infection without neutropenia (Infections and infestations) | 6 (18)
Infection/Febrile Neutropenia-Other (Specify, infection: other:viral; infection: sinusitis) (Infections and infestations) | 2 (3)
Lymphatics (Blood and lymphatic system disorders) | 2 (2)
Lymphatics-Other (Specify, lymphedema) (Blood and lymphatic system disorders) | 1 (1)
Bicarbonate (Metabolism and nutrition disorders) | 4 (7)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (49)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 4 (5)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (45)
Hypokalemia (Metabolism and nutrition disorders) | 10 (19)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (20)
Hyponatremia (Metabolism and nutrition disorders) | 10 (32)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (17)
Musculoskeletal-Other (Specify, pain other: tenderness at catheter site; pain: cathether placement) (Metabolism and nutrition disorders) | 1 (1) — pain: musculoskeletal LT forearm RUE; r/t phlebitis
Dizziness/lightheadedness (Nervous system disorders) | 3 (3)
Insomnia (Nervous system disorders) | 1 (1)
Mood alteration-anxiety, agitation (Nervous system disorders) | 1 (2)
Mood alteration-depression (Nervous system disorders) | 3 (3)
Neuropathy-sensory (Nervous system disorders) | 4 (4)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Keratitis (corneal inflammation/corneal ulceration) (Eye disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Abdominal pain or cramping (Gastrointestinal disorders) | 2 (3)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (9)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 4 (6)
Pain-Other (Specify, Pain Other: tenderness at catheter site) (General disorders) | 4 (5) — Pain: catheter placement Pain: musculoskeletal LT forearm RUE; r/t phlebitis Bone pain
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pulmonary-Other (Specify, Pulmonary Other: bronchospasm/wheezing) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine (Renal and urinary disorders) | 1 (2)
Dysuria (painful urination) (Renal and urinary disorders) | 4 (4)
Incontinence (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 6 (17)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (3)
Urine color change (not related to other dietary or physiologic cause e.g., bilirubin, concentrated (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed to accrual due to very poor enrollment. No meaningful data analysis was possible on the small number of accrued subjects, so none was done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No